CLINICAL TRIAL: NCT05508958
Title: Optimising Recovery After Cup Revision - is the Anterior Approach Superior to Posterolateral?
Brief Title: Cup Revisions Through Anterior or Posterolateral Approach: an RCT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Reinier Haga Orthopedisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OC-2020-018
Record Dates: First submitted 2022-08-12; First posted 2022-08-19 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Loosening, Prosthesis
Keywords: Isolated cup revision; Hip revision surgery; Anterior approach; Posterolateral approach; Cup revision surgery
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Physiotherapist assessing functional tests will be blinded for treatment. Data analyst will be blinded for treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior approach (Experimental): Cup revision surgery through the anterior approach
  Interventions: Procedure: Anterior approach
- Posterolateral approach (Active Comparator): Cup revision surgery through the posterolateral approach
  Interventions: Procedure: Posterolateral approach

INTERVENTIONS:
Procedure: Anterior approach — Anterior approach
  Arms: Anterior approach
Procedure: Posterolateral approach — Posterolateral approach
  Arms: Posterolateral approach

SUMMARY:
With increasing numbers of total hip arthroplasties performed each year, the incidence of problems related to loosening and wear of total hip arthroplasties is expected to also increase. While the anterior approach for primary total hip arthroplasty has demonstrated to result in a faster short-term recovery than the traditional lateral and posterior approach, this effect has not yet been investigated in revision surgery. Accelerating functional outcome may increase patient satisfaction and reduce healthcare costs.

The primary objective is to assess whether isolated cup revision surgery through the anterior approach results in increased functional status and higher patient satisfaction than through the posterolateral approach.

This is a prospective Randomized Controlled Trial (RCT) in which 68 patients will be included (34 per group). Patients will be evaluated preoperatively and 6 weeks, 3 months and 1 year postoperatively.

The main endpoints are functional recovery as measured with the 30-sec Chair Stand Test (30s-CST), 40m Fast Paced Walking Test (40m FPWT) and the Stair Climb Test (SCT).

Secondary endpoints are Modified Borg scale outcomes after the functional tests, Numeric Rating Scale (NRS) for pain (rest/movement), Oxford Hip Score (OHS), HOOS-PS, EQ-5D-5L, satisfaction, cup inclination and complications at 30 days and 90 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* On waiting list or scheduled for isolated cup revision surgery through anterior or posterolateral approach
* A good command of the Dutch language

Exclusion Criteria:

* Revision for confirmed or suspected infection
* Not suitable for both approaches under study, as judged by orthopaedic surgeon
* Unable to fully understand study information and to accurately/reliably complete the questionnaires, as judged by researcher and/or orthopaedic surgeon
* Unable to accurately follow instructions for study procedures / measurements, as judged by researcher and/or orthopaedic surgeon
* Unwilling to sign informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline 30-sec Chair Stand Test (30s-CST) at 6 weeks | 6 weeks postoperatively
  The 30 second Chair Stand Test (30s-CST) is designed to test the sit-to-stand activity, incorporating lower body strength and dynamic balance, and measures the maximum number of chair stand repetitions possible in a 30 second period. It is part of the core set of tests to assess physical function in patients with hip or knee osteoarthritis or following joint arthroplasty, as recommended by the Osteoarthritis Research Society International (OARSI).
Change from baseline 40m Fast Paced Walk Test (40m FPWT) at 6 weeks | 6 weeks postoperatively
  The 40m Fast Paced Walk Test (40m FPWT) tests walking speed over short distances and changing directions during walking. It is timed over 4 x 10 meters, for a total of 40 meters. It is part of the core set of tests to assess physical function in patients with hip or knee osteoarthritis or following joint arthroplasty, as recommended by the Osteoarthritis Research Society International (OARSI).
Change from baseline Stair Climb Test (SCT) at 6 weeks | 6 weeks postoperatively
  The Stair Climb Test (SCT) is designed to test ascending and descending stair activity, and measures the time in seconds to ascend and descend a flight of stairs. It is part of the core set of tests to assess physical function in patients with hip or knee osteoarthritis or following joint arthroplasty, as recommended by the Osteoarthritis Research Society International (OARSI).

SECONDARY OUTCOMES:
Change from baseline Modified Borg Rating of Perceived Exertion (RPE) scale outcome during 30s-CST at 6 weeks, 3 months and 1 year | Preoperatively, and 6 weeks, 3 months and 1 year postoperatively.
  We will use the Borg RPE scale to assess the patients' perception of effort during the functional tasks
Change from Modified Borg Rating of Perceived Exertion (RPE) scale outcome during 40m FPWT at 6 weeks, 3 months and 1 year | Preoperatively, and 6 weeks, 3 months and 1 year postoperatively.
  We will use the Borg RPE scale to assess the patients' perception of effort during the functional tasks
Change from Modified Borg Rating of Perceived Exertion (RPE) scale outcome during SCT at 6 weeks, 3 months and 1 year | Preoperatively, and 6 weeks, 3 months and 1 year postoperatively.
  We will use the Borg RPE scale to assess the patients' perception of effort during the functional tasks
Change from baseline 30-sec Chair Stand Test (30s-CST) at 6 weeks, 3 months and 1 year | Preoperatively, and 6 weeks, 3 months and 1 year postoperatively
  The 30 second Chair Stand Test (30s-CST) is designed to test the sit-to-stand activity, incorporating lower body strength and dynamic balance, and measures the maximum number of chair stand repetitions possible in a 30 second period. It is part of the core set of tests to assess physical function in patients with hip or knee osteoarthritis or following joint arthroplasty, as recommended by the Osteoarthritis Research Society International (OARSI).
Change from baseline 40m Fast Paced Walk Test (40m FPWT) at 6 weeks, 3 months and 1 year | Preoperatively, and 6 weeks, 3 months and 1 year postoperatively
  The 40m Fast Paced Walk Test (40m FPWT) tests walking speed over short distances and changing directions during walking. It is timed over 4 x 10 meters, for a total of 40 meters. It is part of the core set of tests to assess physical function in patients with hip or knee osteoarthritis or following joint arthroplasty, as recommended by the Osteoarthritis Research Society International (OARSI).
Change from baseline Stair Climb Test (SCT) at 6 weeks, 3 months and 1 year | Preoperatively, and 6 weeks, 3 months and 1 year postoperatively
  The Stair Climb Test (SCT) is designed to test ascending and descending stair activity, and measures the time in seconds to ascend and descend a flight of stairs. It is part of the core set of tests to assess physical function in patients with hip or knee osteoarthritis or following joint arthroplasty, as recommended by the Osteoarthritis Research Society International (OARSI).
Patient reported outcome measure: Pain at rest | Preoperatively, and 6 weeks, 3 months and 1 year postoperatively.
  Measured using Numeric Rating Scale (NRS) for pain at rest
Patient reported outcome measure: Pain during movement | Preoperatively, and 6 weeks, 3 months and 1 year postoperatively.
  Measured using Numeric Rating Scale (NRS) for pain during movement
Patient reported outcome measure: Oxford Hip Score (OHS) | Preoperatively, and 6 weeks, 3 months and 1 year postoperatively.
  The Oxford Hip Score (OHS) is a hip specific questionnaire, consisting of 12 items concerning pain and daily functions. In the original scoring, each question is scored on a 5-point Likert scale, ranging from 1 (no pain/easy to do) to 5 (unbearable/impossible to do). The original total score ranges from 12 (best) to 60 (worst) points. It has been developed for total hip surgery. In the revised scoring, each question is scored from 0 (worst) to 4 (best), ranging the total score from 0 (worst) to 48 (best) (20). The revised scoring will be used in this study.
Patient reported outcome measure: HOOS-PS | Preoperatively, and 6 weeks, 3 months and 1 year postoperatively.
  The HOOS-PS is a short measure of physical function for hip osteoarthritis (OA), derived from the original, longer, Hip disability and Osteoarthritis Outcome Score (HOOS). The raw scoring ranges from 0 (none) to 4 (extreme) per question, for a total raw score range of 0 to 20 (lower is less difficulty). The person interval level score ranges, which can be calculated from the total raw score using a nomogram, ranges from 0 (no difficulty) to 100 (extreme difficulty).
Patient reported outcome measure: EQ-5D-5L | Preoperatively, and 6 weeks, 3 months and 1 year postoperatively.
  EuroQol-5D (EQ-5D) is a general health-related quality of life questionnaire and consists of five questions regarding mobility, self-care, usual activities, pain/discomfort and anxiety/depression and one visual analog scale (VAS) to document the perceived quality of life. It is also used to assess quality adjusted life years (QALY).
Patient reported outcome measure: Satisfaction | 6 weeks, 3 months and 1 year postoperatively.
  Anchor question regarding how satisfied the subject is (in general) with the results of his/her hip surgery?
Cup inclination | 6 weeks postoperatively
  Categorized into ≤35°, 35° - 45° and ≥45°
Complications | 30 days postoperatively and 90 days postoperatively
  Postoperative complications as recorded in the electronic patient file

OTHER OUTCOMES:
Lowgrade infection | 6 weeks, 3 months and 1 year postoperatively.
  To investigate selection bias caused by loss to follow up, the investigators will also record whether a lowgrade infection was determined during or after revision surgery.

CONTACTS AND LOCATIONS:
Overall Officials: M. Rutgers, MD, Principal Investigator — Reinier Haga Orthopedisch Centrum
Locations (1):
- Reinier Haga Orthopedic Center, Zoetermeer, Netherlands